CLINICAL TRIAL: NCT06439121
Title: Effect of the 4-7-8 Breathing Technique on Pain and Nausea-Vomiting in Patients After Bariatric Surgery
Brief Title: The 4-7-8 Breathing Technique on Pain and Nausea-Vomiting
Acronym: Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Eda Özyürek, Ankara Yildirim Beyazıt University, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PAINVOMIT
Record Dates: First submitted 2024-05-13; First posted 2024-06-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pain; Vomiting; Nausea; Post Operative Pain; Vomiting, Postoperative; Nausea, Postoperative
MeSH Terms: conditions — Pain; Vomiting; Nausea; Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-7-8 Breathing Technique (Experimental): The Patient Introduction Form comprises three sections. The first section covers sociodemographic characteristics, including gender, age, BMI, education level, smoking status, and family history of obesity (6 questions). The second section addresses medical characteristics such as chronic diseases, ASA score, duration of general anesthesia, type of surgery, surgical complications history, and length of hospital stay (7 questions).
  The third section evaluates pain and nausea-vomiting using the Visual Analog Scale, a 10 cm horizontal line where patients mark their severity level. Scores range from 0-10, with higher scores indicating increased symptom severity. The scale is versatile, assessing symptoms like pain, anxiety, fatigue, and nausea-vomiting, with vomiting assessed as "present" or "absent." Patients will be taught the 4-7-8 breathing technique pre-surgery and asked to practice it post-surgery. Their responses to the third section's questions will be recorded.
  Interventions: Procedure: 4-7-8 Breathing Technique
- Control (No Intervention): The Patient Introduction Form comprises three sections:
  1. Sociodemographic characteristics, encompassing gender, age, BMI, education level, smoking status, and family history of obesity (6 questions).
  2. Medical characteristics, including the presence of chronic diseases, ASA score, duration of general anesthesia, type of surgery performed, history of surgical complications, and length of hospital stay (7 questions).
  3. Evaluation of pain and nausea-vomiting using the Visual Analog Scale, which entails a 10 cm horizontal line where patients mark their severity level. Scores range from 0-10, with higher scores indicating increased symptom severity. Vomiting will be assessed as "present" or "absent." Patients in the control group will undergo routine monitoring and treatments without interventions, and their responses to the questions from the third section will be recorded.

INTERVENTIONS:
Procedure: 4-7-8 Breathing Technique — Patients will be instructed to practice the 4-7-8 breathing technique once per hour (4 breaths) post-surgery. Pain and nausea-vomiting will be monitored at 0, 2, 6, 12, and 24 hours during their 24-hour hospital stay.
  Arms: 4-7-8 Breathing Technique

SUMMARY:
This study is planned as a randomized controlled trial to determine the effect of the 4-7-8 breathing technique applied to patients after bariatric surgery on pain and nausea and vomiting. The research will be conducted on 60 patients who underwent bariatric surgery between 05.2024-12.2024.

Randomization will be ensured for students who meet the inclusion criteria, and they will be divided into two random groups: the experimental group (n=30) and the control group (n=30). After obtaining consent with the "Informed Consent Form," patients who agree to participate in the study will have the "Patient Introduction Form" filled out by researchers, and they will be provided with training on the 4-7-8 breathing technique. Patients will be instructed to practice the 4-7-8 breathing technique once per hour (4 breaths) post-surgery. Pain and nausea-vomiting will be monitored at 0, 2, 6, 12, and 24 hours during their 24-hour hospital stay. The control group, after consenting with the "Informed Consent Form" the day before surgery, will have the "Patient Introduction Form" filled out by researchers, and their pain and nausea-vomiting status will be monitored at the same intervals during their hospital stay. No interventions will be made for the control group; they will receive routine nursing care during their hospital stay.

DETAILED DESCRIPTION:
Obesity is a significant health issue globally, ranking second among preventable causes of death (Güven, Akyolcu 2020). According to the World Health Organization (WHO) data for 2022, more than 2.5 billion adults are overweight, and 890 million are obese. It is known that 43% of adults (43% of men and 44% of women) are overweight (WHO, 2022). The severity of the situation in Turkey is highlighted in the World Health Organization report, where Turkey ranks first in Europe with a 32% obesity rate (WHO European Regional Obesity Report 2022).

Obesity increases the risk of life-threatening diseases and chronic conditions (WHO, 2006). In 2019, an estimated 5 million deaths occurred due to diseases caused by obesity, such as cardiovascular diseases, diabetes, cancers, neurological disorders, chronic respiratory diseases, and digestive disorders (Collaborators, G. B. D., & Ärnlöv, 2020).

Bariatric surgery is considered the most effective and permanent method for weight loss in obesity treatment (Güngör 2012). The role of nurses is crucial in preventing complications after bariatric surgery (cardiopulmonary complications, venous thromboembolism, anastomotic leakage, electrolyte imbalance) and providing appropriate care when complications occur. Additionally, nurses play a key role in other important aspects of care after bariatric surgery, such as pain management, wound care, drain monitoring, early mobilization, fluid monitoring, nutrition, nausea-vomiting monitoring, continuous education, and psychosocial support (Yılmaz Güven, Arık, Çelik 2021).

Pain caused by tissue damage in bariatric surgery patients, considered the fifth vital sign, should be carefully evaluated and recorded (Berk Özcan 2021). In a study by Steyer et al., it was found that nurses most commonly diagnosed pain in patients undergoing bariatric surgery (Steyer et al., 2016). Surgical pain that interferes with patients' physical movement and daily life activities can prolong the recovery process and lead to complications. Therefore, it is important to regularly assess pain levels with pain scales within the first 24 hours after surgery and manage pain accordingly (Usta 2014; Schulman and Thompson 2017). Postoperative nausea and vomiting in patients due to surgical intervention and anesthesia continue to be a common problem (Grindel and Grindel 2006; Varner KL, March AL 2020). Horizontal resection of the stomach, pressure applied by stapling and suturing lines to the stomach tissue, and the pressure applied to the abdomen by insufflation with CO2 during laparoscopic procedures in bariatric surgery increase the risk of postoperative nausea-vomiting (Aftab et al. 2019; Kushner et al. 2020). Post-bariatric surgery, especially within the first 24 hours, nausea and vomiting can be observed in 65% of patients (Ruhaiyem et al. 2016). The importance of performing correct and regular breathing exercises to minimize these problems is significant. Upon reviewing the literature, it is observed that there are a limited number of studies using the 4-7-8 Breathing Technique after bariatric surgery (Kurt Aktaş, Eskici İlgin 2023; Eskici İlgin, Yayla 2023). In one study, it was observed that the 4-7-8 Breathing Technique reduced the anxiety levels of patients after bariatric surgery (Kurt Aktaş, Eskici İlgin 2023). In another study, it was determined that the 4-7-8 breathing exercise reduced post-laparoscopic bariatric surgery pain and improved sleep quality (Eskici İlgin, Yayla 2023).

Materials and Methods Study Design This research will be conducted using an experimental research model to determine the effect of the 4-7-8 breathing technique on pain and nausea-vomiting in patients after bariatric surgery.

Population and Sample of the Study The population of the study will consist of patients who will undergo bariatric surgery admitted to the General Surgery Clinic of T.C. Ministry of Health Etlik City Hospital. There are 11 nurses working in the General Surgery Clinic where the research will be conducted, and it has a capacity of 22 beds.

The sample of the study will consist of patients who underwent bariatric surgery between May 2024 and October 2024 and meet the criteria for participation in the study.

The sample size was calculated using the G-power 3.1 program before the study, and based on the data of Doğan and Arslan (2022), with 80% power, 0.05 error, and 0.30 effect size, the sample size was determined as 46 patients. Considering the possibility of missing data, the sample will be increased by 30%, and thus, 60 patients will be included in the study.

Patients who meet the research criteria will be assigned to the experimental and control groups in a 1:1 ratio by block randomization, using a computer program-generated (https://www.random.org) sequence.

Inclusion criteria for the study: Being 18 years of age and older, and under 65 years of age, Undergoing laparoscopic general surgery under general anesthesia (such as laparoscopic sleeve gastrectomy, Laparoscopic Roux-en-Y gastric bypass), Being ASA Score I or II, Being willing to participate in the study Exclusion criteria for the study: Not undergoing laparoscopic surgical intervention, Having neurological or psychological problems, Transferred to the intensive care unit after surgery, Emergency and unplanned cases, Patients diagnosed with cancer will be excluded from the study.

Data Collection Tools The patient identification form will be used to collect research data. This form consists of 3 sections. The first section will include sociodemographic characteristics consisting of 6 questions, including gender, age, BMI, education level, smoking status, and family history of obesity.

The second section will include medical characteristics consisting of 7 questions, including the presence of chronic disease, ASA score, duration of stay under general anesthesia, type of surgery performed, history of surgical complications, and length of hospital stay.

The third section will include 3 questions to evaluate pain and nausea-vomiting. Visual analog scale will be used to evaluate pain and nausea. The scale consists of a horizontal line 10 cm in length, and the distance between the far left end of the scale and the point marked by the patient determines the score. The score range from this scale is between 0-10, and higher scores indicate increased severity of the symptoms being evaluated. This scale can be used to evaluate various symptoms such as pain, anxiety, fatigue, nausea, vomiting. Vomiting will be evaluated as "present" or "absent".

Ethics of the Study Permission obtained from the Ankara Yıldırım Beyazıt University Ethics Committee and the management of Etlik City Hospital where the study will be conducted. Patients will be informed about the research and their consent will be obtained.

Data Evaluation IBM SPSS Statistics 23.0 software will be used for statistical analysis and calculations. Frequency distribution (number, percentage) will be provided for categorical variables, and descriptive statistics (mean, standard deviation) will be provided for numerical variables during data evaluation. The normal distribution status of the data will be evaluated using the Shapiro-Wilk test. In cases where the data does not follow a normal distribution, the Mann Whitney-U test and Spearman correlation analysis will be used to determine differences between the two groups. A significance level of p<0.05 will be accepted.

Data Collection For the experimental group, after obtaining permission with the "Informed Consent Form" the day before surgery, patients who agree to participate in the research will be provided with a "Patient Introduction Form" and will be given training on the 4-7-8 breathing technique. Patients will be instructed to apply the 4-7-8 breathing technique as 1 set (4 breaths) per hour after surgery. Pain and nausea-vomiting status will be monitored at 0, 2, 6, 12, and 24 hours during the 24-hour period of hospitalization.

Holding the breath for a period helps renew the body's oxygen. The 4-7-8 breathing technique provides the oxygen support needed by organs and tissues and helps to expel CO2. In the 4-7-8 breathing technique, a breath is taken for 4 seconds, held for 7 seconds, and exhaled in 8 seconds (How to use the 4-7-8 breathing technique to reduce stress https://www.medicalnewstoday.com/articles/324417. March 22, 2024).

For the control group, after obtaining permission with the "Informed Consent Form" the day before surgery, patients who agree to participate in the research will be provided with a "Patient Introduction Form". Pain and nausea-vomiting status will be monitored at 0, 2, 6, 12, and 24 hours during the 24-hour period of hospitalization. No intervention will be made for patients in the control group, and they will receive routine nursing care provided at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 and above, and under 65 years old
* Patients undergoing laparoscopic general surgery under general anesthesia (such as laparoscopic sleeve gastrectomy, Laparoscopic Roux-en-Y gastric bypass) will be included in the study.
* Having an ASA Score of I or II
* Being willing to participate in the study

Exclusion Criteria:

* Not undergoing laparoscopic surgical intervention,
* Having neurological or psychological issues,
* Transferred to the intensive care unit after surgery,
* Emergency and unplanned cases,
* Patients diagnosed with cancer will be excluded from the scope of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Pain Scale | just before operation, just after operation
  During the 24-hour hospital stay, the patient's pain level will be assessed at 0, 2, 6, 12, and 24 hours, and the pain intensity, ranging from 0 for no pain to 10 for severe pain, as indicated by the patient, will be recorded.
Vomitting | just before operation, just after operation
  During the 24-hour hospital stay, the patient's nausea level will be observed at 0, 2, 6, 12, and 24 hours, and the occurrence of vomiting, noted as either present or absent, will be recorded.
Nausea | just before operation, just after operation
  During the 24-hour hospital stay, the patient's nausea level will be assessed at 0, 2, 6, 12, and 24 hours, and the severity of nausea, ranging from 0 for no nausea to 10 for severe nausea as indicated by the patient, will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara YBU, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No